CLINICAL TRIAL: NCT04186624
Title: Effectiveness of Supervised Exercise Program After Subacromial- Subdeltoid Bursitis Injection in Subacromial Impingement Syndrome
Brief Title: Effectiveness of Supervised Exercise Program in Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Kardelen Gencer Atalay, Principal Investigator, Marmara University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2019.347
Record Dates: First submitted 2019-11-25; First posted 2019-12-05 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-02

CONDITIONS: Subacromial Impingement Syndrome
Keywords: Subacromial Impingement Syndrome; Subacromial-subdeltoid bursa corticosteroid injection; Exercise Therapy
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Intervention Model Description: This randomized controlled study is designed to have two groups with a single arm.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supervised Exercise Program (Experimental): The exercise program that applied at the hospital includes rotator cuff and scapular muscle strengthening, stretching and active-assistive range of motion exercises and proprioceptive neuromuscular facilitation exercises.
  Interventions: Drug: Subacromial-subdeltoid bursa corticosteroid injection
- Home-based Exercise Program (Active Comparator): The home-based exercise program given with a brochure that includes rotator cuff and scapular muscle strengthening, stretching and active-assistive range of motion exercises and proprioceptive neuromuscular facilitation exercises.
  Interventions: Drug: Subacromial-subdeltoid bursa corticosteroid injection

INTERVENTIONS:
Drug: Subacromial-subdeltoid bursa corticosteroid injection — 1 ml (7 mg / ml) betamethasone and 4 ml of 0.5% bupivacaine will be given subacromial bursa-subdeltoid space. Injection will be performed ultrasound-guided while the patient is in sitting position with the lateral approach.
  Other Names: Subacromial-subdeltoid bursa injection

SUMMARY:
Subacromial Impingement Syndrome (SIS) is a pathology resulting from mechanical repetitive compression and inflammation of the supraspinatus tendon, subacromial bursa and biceps tendon under the acromion and the coracoacromial ligament. It is the most common cause of shoulder pain, with an incidence of 44-65%. Restriction of the range of motion, along with the pain in the anterior region of the shoulder, is the main reason for disability and decreased quality of life in patients with SIS. Physical exercises to improve the range of motion, strengthening, and flexibility is the main part of treatment. The subacromial-subdeltoid bursa corticosteroid injection is shown to decrease pain during the exercise program and increase participation in the treatment. This study aims to compare the effectiveness of a supervised exercise program and home-based exercise program after subacromial-subdeltoid bursa corticosteroid injection in patients with SIS.

DETAILED DESCRIPTION:
Subacromial Impingement Syndrome (SIS) is a pathology resulting from mechanical repetitive compression and inflammation of the supraspinatus tendon, subacromial bursa and biceps tendon under the acromion and the coracoacromial ligament. It was first described in 1972 by Neer. Neer described SIS as a progressive syndrome with three stages, beginning with chronic bursitis and proceeding to partial and complete tears of the supraspinatus tendon, which may extend to rupture of other parts of the rotator cuff and may also involve the long biceps tendon. SIS is one of the most common causes of shoulder pain and disability reasons in both primary and secondary care. It is characterized by functional impairment of shoulder resulted from the progressive limitation of both active and passive glenohumeral movements. Restriction of the range of motion (ROM) along with the pain in the anterior region of the shoulder that gets worse with arm elevation or overhead activities is the main reason for decreased quality of life in patients with SIS. Therapeutic exercise programs are commonly used treatment methods in relieving pain and improving ROM and muscle elasticity. It was shown that such programs are more effective in reducing pain and improving functional loss than placebo in both short- and long-term. However, the optimal exercise regimen with the variety, frequency, and intensity exercises is still unclear. It is also controversial if a supervised exercise program is superior to a prescribed home-based exercise program. An efficient exercise program should target all structures affected by subacromial impingement. Therefore, both supervised and home-based exercise programs must involve rotator cuff and scapular stabilizing muscle strengthening, stretching and active-assistive range of motion exercises and proprioceptive neuromuscular facilitation exercises. Corticosteroid injection into the subacromial-subdeltoid bursa is shown to increase participation, decrease pain during the exercise program, and found to be effective for symptomatic impingement. The analgesic effect provides significant improvement of functions mainly in the short-term. Therefore, some physicians prefer corticosteroid injections alone in the treatment of SIS. However, it was found that the combination of corticosteroid injection and exercise program is significantly superior to corticosteroid injections alone. Ultrasound-guided subacromial-subdeltoid bursa injections are shown to have better outcome results than blind injections for both pain and overall shoulder function. This study aims to compare the effectiveness of supervised exercise and home-based exercise programs after ultrasound-guided subacromial-subdeltoid bursa corticosteroid injection in patients with SIS.

Patients diagnosed with SIS will be included and randomized into two groups. Both groups will receive subacromial-subdeltoid bursa 1 ml (7 mg/ml) betamethasone and 4 ml of 0.5% bupivacaine injection. The injection will be performed ultrasound-guided while the patient is in a sitting position with the lateral approach. The first group will perform their exercises under the supervision of the physiotherapist in the hospital. The second group will be taken to the home-based exercise program in a brochure format. Thus, both groups will receive the same exercises every day.

The pain will be assessed with the Visual Analogue Scale (VAS), active and passive ROM will be measured with a goniometer before injection, immediately, first hour, third week, and third month after the injection. The quality of life will be evaluated by Short Form 36, and disability will be questioned by Shoulder Pain and Disability Index before injection and third week and third month after injection.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms lasting longer than 3 months
2. Aged between 20-60 years
3. The diagnosis is made by the clinician and detected by MRI

Exclusion Criteria:

1. History of physical therapy or injection in the last 3 months
2. Shoulder fracture history
3. Presence of Type III (hooked) acromion
4. Complete rupture of the rotator cuff muscles
5. Presence of instability problem in shoulder
6. History of shoulder surgery
7. History of inflammatory rheumatoid disease
8. Uncontrolled diabetes mellitus
9. Allergy to steroids or local anesthetics (drug hypersensitivity)
10. Known contraindications for interventional procedures (infection at the injection site, coagulopathy, etc.)

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Pain and tightness sensation | before treatment (T0)
  Shoulder pain and sensations of tightness will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable)
Pain and tightness sensation | 1st hour after injection (T1)
  Shoulder pain and sensations of tightness will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable)
Pain and tightness sensation | 3rd week of treatment (T2)
  Shoulder pain and sensations of tightness will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable)
Pain and tightness sensation | 3rd month of treatment (T3)
  Shoulder pain and sensations of tightness will be evaluated with a 10-cm horizontal visual analogue scale (VAS) ranging from "0 cm" (no discomfort) to "10 cm" (worst imaginable)

SECONDARY OUTCOMES:
Pain and Disability - SPADI | before treatment (T0)
  Shoulder Pain and Disability Index (SPADI) is a questionnaire developed to assess pain and disability related to shoulder problems. Pain dimension has 5 questions regarding the pain severity. Functional activities are assessed with 8 questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. Each question is scored between 0 and 10, and high scores indicate increased severity and high scores indicate increased severity (0 = no difficulty and 10 = so difficult it require help) .The validity and reliability of the questionnaire in Turkish were conducted by Bumin et al.
Pain and Disability - SPADI | 3rd week of treatment (T1)
  Shoulder Pain and Disability Index (SPADI) is a questionnaire developed to assess pain and disability related to shoulder problems. Pain dimension has 5 questions regarding the pain severity. Functional activities are assessed with 8 questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. Each question is scored between 0 and 10, and high scores indicate increased severity and high scores indicate increased severity (0 = no difficulty and 10 = so difficult it require help) .The validity and reliability of the questionnaire in Turkish were conducted by Bumin et al.
Pain and Disability - SPADI | 3rd month of treatment (T2)
  Shoulder Pain and Disability Index (SPADI) is a questionnaire developed to assess pain and disability related to shoulder problems. Pain dimension has 5 questions regarding the pain severity. Functional activities are assessed with 8 questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. Each question is scored between 0 and 10, and high scores indicate increased severity and high scores indicate increased severity (0 = no difficulty and 10 = so difficult it require help) .The validity and reliability of the questionnaire in Turkish were conducted by Bumin et al.
Quality of life- Short Form-36 | before treatment (T0)
  Short Form-36 (SF-36) is a widely-used and well-documented health-related quality of life index. The SF-36 consists of 36 questions; It survey has eight sub-dimensions, including physical functioning, role limitations due to physical problems, pain, general health perception, mental health, role limitations due to emotional problems, vitality, and social functioning, which are evaluated individually. A higher score on a 0-100 scale indicates a better quality of life.
Quality of life- Short Form-36 | 3rd week of treatment (T1)
  Short Form-36 (SF-36) is a widely-used and well-documented health-related quality of life index. The SF-36 consists of 36 questions; It survey has eight sub-dimensions, including physical functioning, role limitations due to physical problems, pain, general health perception, mental health, role limitations due to emotional problems, vitality, and social functioning, which are evaluated individually. A higher score on a 0-100 scale indicates a better quality of life.
Quality of life- Short Form-36 | 3rd month of treatment (T2)
  Short Form-36 (SF-36) is a widely-used and well-documented health-related quality of life index. The SF-36 consists of 36 questions; It survey has eight sub-dimensions, including physical functioning, role limitations due to physical problems, pain, general health perception, mental health, role limitations due to emotional problems, vitality, and social functioning, which are evaluated individually. A higher score on a 0-100 scale indicates a better quality of life.
Shoulder range of motion (ROM) will be evaluated with a goniometer | before treatment (T0)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, internal and external rotation.
Shoulder range of motion (ROM) will be evaluated with a goniometer | 1st hour after injection (T1)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, internal and external rotation.
Shoulder range of motion (ROM) will be evaluated with a goniometer | 3rd week of treatment (T2)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, internal and external rotation.
Shoulder range of motion (ROM) will be evaluated with a goniometer | 3rd month of treatment (T3)
  Shoulder range of motion (ROM) will be evaluated with a goniometer in all directions; flexion, extension, abduction, internal and external rotation.

CONTACTS AND LOCATIONS:
Overall Officials: İlker Yağcı, Prof, Study Chair — Marmara University; Ebru Kaplan, PT, Principal Investigator — Marmara University
Locations (1):
- Marmara University School of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pieters L, Lewis J, Kuppens K, Jochems J, Bruijstens T, Joossens L, Struyf F. An Update of Systematic Reviews Examining the Effectiveness of Conservative Physical Therapy Interventions for Subacromial Shoulder Pain. J Orthop Sports Phys Ther. 2020 Mar;50(3):131-141. doi: 10.2519/jospt.2020.8498. Epub 2019 Nov 15. PMID 31726927
- [Background] Granviken F, Vasseljen O. Home exercises and supervised exercises are similarly effective for people with subacromial impingement: a randomised trial. J Physiother. 2015 Jul;61(3):135-41. doi: 10.1016/j.jphys.2015.05.014. Epub 2015 Jun 18. PMID 26093810
- [Background] Steuri R, Sattelmayer M, Elsig S, Kolly C, Tal A, Taeymans J, Hilfiker R. Effectiveness of conservative interventions including exercise, manual therapy and medical management in adults with shoulder impingement: a systematic review and meta-analysis of RCTs. Br J Sports Med. 2017 Sep;51(18):1340-1347. doi: 10.1136/bjsports-2016-096515. Epub 2017 Jun 19. PMID 28630217
- [Background] Burger M, Africa C, Droomer K, Norman A, Pheiffe C, Gericke A, Samsodien A, Miszewski N. Effect of corticosteroid injections versus physiotherapy on pain, shoulder range of motion and shoulder function in patients with subacromial impingement syndrome: A systematic review and meta-analysis. S Afr J Physiother. 2016 Sep 27;72(1):318. doi: 10.4102/sajp.v72i1.318. eCollection 2016. PMID 30135893
- [Background] Kromer TO, de Bie RA, Bastiaenen CH. Effectiveness of physiotherapy and costs in patients with clinical signs of shoulder impingement syndrome: One-year follow-up of a randomized controlled trial. J Rehabil Med. 2014 Nov;46(10):1029-36. doi: 10.2340/16501977-1867. PMID 25211291